## ID:2014-027

## **Dexmedetomidine-ketamine in Femur Proximal Fracture Patients**

## NCT02150759

## 04-24-2019

This study was approved by the institutional review board of Inje University Haeundae Paik Hospital (129792-2014-027) and written informed consent was obtained from patients. This study was registered before patient enrollment began at ClinicalTrials.gov (NCT02150759; date of registration: December 23, 2013).

We hypothesized that ketamine or fentanyl could be better analgesics to control movement evoked pain in elderly patients with proximal femur fracture who were undergoing DEX continuous infusion.

We compared the analgesic effect of Dexmedetomidine (1mcg/kg)- fentanyl (1mcg/kg) combination vs dexmedetomidine (1mcg/kg) - ketantire (1mg/kg) combination. After 10 minutes of drug infusion, patients are prepared for spiral anesthesia. Pain scale and quality of patient during lateral positioning for spinal anesthesia were measured three times (lateral position, chest-knee position, intrathecal local anesthetics injection)

Pain score (0 = calm, 1 = facial grinaring, 2 = moaning 3 = screaming, 4 = unable to proceed because of restlessness of agrication) of patient position maintained for spinal block was recorded. Quality score (0 = not satisfactory, 1 = prisfactory, 2 = good, and 3 = optimal) of patient position maintained for spinal block was recorded. Data are presented as the number of patients.

Data were analyzed using Medcalc 14.12.0 (MedCalc Software bvba, Ostend, Belgium). Parametric variables were described as mean  $\pm$  standard deviation (SD). Qualitative variables were described as number and as median (interquartile range). Student's t-test, Fisher's exact test, or Mann-Whitney U-test was used as appropriate to compare the two groups. P < 0.05 was considered to indicate strainical significant.